CLINICAL TRIAL: NCT00756977
Title: BLI850 vs an Active Control Bowel Preparation in Adult Subjects Undergoing Colonoscopy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Braintree Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BLI850-301; BLI850-301
Record Dates: First submitted 2008-09-18; First posted 2008-09-22 (Estimated); Results first posted 2013-08-09 (Estimated); Last update posted 2013-08-15 (Estimated); Status verified 2013-08

CONDITIONS: Colon Cancer
Keywords: Colonoscopy; screening
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): multi-dose preparation for oral administration prior to colonoscopy
  Interventions: Drug: BLI850
- 2 (Active Comparator): multi-dose preparation for oral administration prior to colonoscopy
  Interventions: Drug: polyethylene glycol 3350 based bowel preparation

INTERVENTIONS:
Drug: BLI850 — multi-dose preparation for oral administration prior to colonoscopy
  Arms: 1
Drug: polyethylene glycol 3350 based bowel preparation — multi-dose preparation for oral administration prior to colonoscopy
  Arms: 2

SUMMARY:
This is a randomized, parallel, multi-center, single-blind study, comparing BLI850 to an FDA approved bowel preparation in adult subjects undergoing colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female outpatients who are undergoing colonoscopy for a routinely accepted indication, including:

   * Evaluation of barium enema results
   * GI bleeding
   * Anemia of unknown etiology
   * Neoplastic disease surveillance
   * Abnormal Endosonography
   * Inflammatory bowel disease
   * Unknown diarrhea or constipation etiology
   * Polypectomy
   * Laser therapy
   * Routine screening
2. At least 18 years of age.
3. Otherwise in good health, as determined by physical exam and medical history.
4. If female, and of child-bearing potential, is using an acceptable form of birth control (hormonal birth control, IUD, double-barrier method, depot contraceptive, abstinent, or vasectomized spouse).
5. Negative urine pregnancy test at screening, if applicable.
6. In the Investigator's judgment, subject is mentally competent to provide informed consent to participate in the study.

Exclusion Criteria:

1. Subjects with known or suspected ileus, severe ulcerative colitis, gastrointestinal obstruction, gastric retention, bowel perforation, toxic colitis, or megacolon.
2. Subjects with impaired consciousness that predisposes them to pulmonary aspiration.
3. Subjects who are undergoing colonoscopy for foreign body removal or decompression.
4. Subjects with clinically significant electrolyte abnormalities based on Visit 1 laboratory results.
5. Subjects who had previous significant gastrointestinal surgeries (e.g. colostomy, colectomy, gastric bypass).
6. Subjects who are pregnant or lactating, or intending to become pregnant during the study.
7. Subjects of childbearing potential who refuse a pregnancy test.
8. Subjects who are allergic to any preparation components
9. Subjects who, in the opinion of the Investigator, should not be included in the study for any reason, including inability to follow study procedures.
10. Subjects who have participated in an investigational surgical, drug, or device study within the past 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 394 (Actual)
Dates: Start 2008-08; Primary Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John D McGowan, Study Director — Braintree Laboratories
Locations (12):
- United States (12):
  - University of South Alabama, Mobile, Alabama
  - Jupiter Research, Jupiter, Florida
  - Miami Research Associates, Miami, Florida
  - United Medical Research, New Smyrna Beach, Florida
  - Atlanta Gastroenterology Associates, Roswell, Georgia
  - Delta Research Partners, Monroe, Louisiana
  - Maryland Digestive Disease Research, Laurel, Maryland
  - Long Island GI Research Group, Great Neck, New York
  - Carolina Digestive Health Associates, Harrisburg, North Carolina
  - Wake Research Associates, Raleigh, North Carolina
  - Regional Gastroenterology Associates of Lancaster, Lancaster, Pennsylvania
  - Southeastern Clinical Research, Chattanooga, Tennessee

RESULTS

PARTICIPANT FLOW:
Groups:
- BLI850; Polyethylene Glycol 3350 Based Bowel Preparation: Single administration oral preparation
Period: Overall Study
Arm/Group | BLI850 | Polyethylene Glycol 3350 Based Bowel Preparation
Started | 196 | 198
Completed | 175 | 187
Not Completed | 21 | 11

BASELINE CHARACTERISTICS:
Population: Intent to Treat population
Groups:
- Total: Total of all reporting groups
Arm/Group | BLI850 | Polyethylene Glycol 3350 Based Bowel Preparation | Total
Number analyzed (Participants) | 176 | 190 | 366
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 128 | 141 | 269
  >=65 years | 48 | 49 | 97
Age Continuous [Mean (Standard Deviation); unit: years] | 56.8 (13.1) | 56.9 (12.3) | 56.9 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97 | 104 | 201
  Male | 79 | 86 | 165
Region of Enrollment [Number; unit: participants]
  United States | 176 | 190 | 366

OUTCOME MEASURES:

1. Primary Outcome: Efficacy - Preparation Quality Using a 4 Point Scale
Description: Percentage of patients with a successful preparation (cleaning rated as "Good" or "Excellent"
Time Frame: 2-day
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BLI850 | Polyethylene Glycol 3350 Based Bowel Preparation
Number analyzed (Participants) | 176 | 188
percentage of participants | 90 [84 to 94] | 84 [77 to 89]

2. Secondary Outcome: Serum Chemistry Results (mg/dL)
Description: Change from Baseline
Time Frame: 2 days
Population: Intent-to-treat population: all patients that took any portion of the study preparation.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | BLI850 | Polyethylene Glycol 3350 Based Bowel Preparation
Number analyzed (Participants) | 176 | 190
mg/dL
  Blood urea nitrogen | -3.08 (3.6) | -3.59 (3.9)
  Calcium | -0.08 (0.42) | -0.13 (0.43)
  Creatinine | 0.00 (0.14) | 0.03 (0.12)
  Direct bilirubin | 0.05 (0.05) | 0.05 (0.06)
  Glucose | 0.82 (32) | -5.52 (25)
  Phosphate | -0.08 (0.65) | -0.02 (0.56)
  Total bilirubin | 0.28 (0.21) | 0.27 (0.24)
  Uric acid | 0.39 (0.80) | 0.49 (0.77)

3. Secondary Outcome: Hematology Results (%)
Description: Change from Baseline
Time Frame: 2 days
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: standard %
Arm/Group | BLI850 | Polyethylene Glycol 3350 Based Bowel Preparation
Number analyzed (Participants) | 176 | 190
standard %
  Basophils | 0.03 (0.46) | 0.07 (0.37)
  Eosinophils | 0.06 (0.95) | -0.09 (0.78)
  Hematocrit | 0.50 (3.1) | 0.38 (2.6)
  Lymphocytes | 1.09 (7.3) | 0.44 (6.6)
  Monocytes | -0.05 (1.79) | 0.07 (1.71)
  Neutrophils | -1.08 (8.0) | -0.50 (7.7)

4. Secondary Outcome: Serum Chemistry Results (U/L)
Description: Change from Baseline
Time Frame: 2 days
Population: Intent-to-treat population: all patients that took any portion of the study preparation.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | BLI850 | Polyethylene Glycol 3350 Based Bowel Preparation
Number analyzed (Participants) | 176 | 190
U/L
  Alkaline Phosphatase | 1.46 (10.9) | 1.96 (13.6)
  ALT | 0.93 (8.8) | 4.20 (50.8)
  Amylase | -11.1 (14.7) | -16.5 (97.3)
  AST | 2.63 (6.5) | 2.61 (16.8)
  Creatine kinase | 29.1 (198) | 6.2 (110)
  GGT | -1.38 (11.8) | 0.73 (19.1)

5. Secondary Outcome: Serum Chemistry Results (mEq/L)
Description: Change from Baseline
Time Frame: 2 days
Population: Intent-to-treat population: all patients that took any portion of the study preparation.
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | BLI850 | Polyethylene Glycol 3350 Based Bowel Preparation
Number analyzed (Participants) | 176 | 190
mEq/L
  Anion Gap | 0.71 (2.70) | 0.53 (2.79)
  Bicarbonate | -0.88 (2.6) | -0.51 (2.5)
  Chloride | 0.63 (2.4) | 0.27 (2.4)
  Magnesium | -0.01 (0.13) | -0.03 (0.14)
  Potassium | -0.19 (0.43) | -0.24 (0.46)
  Sodium | 0.47 (2.2) | 0.29 (2.2)

6. Secondary Outcome: Serum Chemistry Results (g/dL)
Description: Change from Baseline
Time Frame: 2 days
Population: Intent-to-treat population: all patients that took any portion of the study preparation.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | BLI850 | Polyethylene Glycol 3350 Based Bowel Preparation
Number analyzed (Participants) | 176 | 190
g/dL
  Albumin | 0.03 (0.23) | -0.00 (0.22)
  Total protein | 0.06 (0.38) | 0.01 (0.36)

7. Secondary Outcome: Serum Chemistry Results (GFR)
Description: Change from Baseline
Time Frame: 2 days
Measure: Mean (Standard Deviation); unit: ml/min
Arm/Group | BLI850 | Polyethylene Glycol 3350 Based Bowel Preparation
Number analyzed (Participants) | 176 | 190
ml/min | -0.21 (14.6) | -2.82 (11.5)

8. Secondary Outcome: Hematology Results (1000/MCL)
Description: Change from Baseline
Time Frame: 2 days
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: 1000/MCL
Arm/Group | BLI850 | Polyethylene Glycol 3350 Based Bowel Preparation
Number analyzed (Participants) | 176 | 190
1000/MCL
  Platelets | 1.82 (36) | -1.09 (36)
  White blood cells | -0.55 (1.6) | -0.59 (1.6)

9. Secondary Outcome: Hematology Results - Hemoglobin
Description: Change from Baseline
Time Frame: 2 days
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | BLI850 | Polyethylene Glycol 3350 Based Bowel Preparation
Number analyzed (Participants) | 176 | 190
g/dL | 0.20 (0.90) | 0.20 (0.75)

10. Secondary Outcome: Hematology Results - Red Blood Cells
Description: Change from Baseline
Time Frame: 2 days
Measure: Mean (Standard Deviation); unit: MILL/MCL
Arm/Group | BLI850 | Polyethylene Glycol 3350 Based Bowel Preparation
Number analyzed (Participants) | 176 | 190
MILL/MCL | 0.07 (0.30) | 0.04 (0.26)

11. Secondary Outcome: Serum Chemistry Results (Osmolality)
Description: Change from Baseline
Time Frame: 2 days
Measure: Mean (Standard Deviation); unit: mOsm/kg
Arm/Group | BLI850 | Polyethylene Glycol 3350 Based Bowel Preparation
Number analyzed (Participants) | 176 | 190
mOsm/kg | -0.88 (6.2) | -0.18 (7.9)

ADVERSE EVENTS:
Time Frame: 2 days
Description: ITT Population - all subjects that took any portion of preparation
Arm/Group | BLI850 | Polyethylene Glycol 3350 Based Bowel Preparation
Serious Adverse Events (participants affected / at risk) | 0/176 | 0/190
Other Adverse Events (participants affected / at risk) | 145/176 | 142/190
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BLI850 (N=176) | Polyethylene Glycol 3350 Based Bowel Preparation (N=190)
abdominal distension (Gastrointestinal disorders) | 92 | 85
abdominal pain (Gastrointestinal disorders) | 71 | 78
nausea (Gastrointestinal disorders) | 74 | 75
overall discomfort (Gastrointestinal disorders) | 122 | 108
vomiting (Gastrointestinal disorders) | 19 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 360 days from the time submitted to the sponsor for review. The sponsor cannot extent the embargo.